CLINICAL TRIAL: NCT05719129
Title: The Stanford Lasting Change Study
Brief Title: The Lasting Change Study
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Snyder, Chair, Dept. of Genetics, Stanford University
Other Study IDs: 66491, 68645
Record Dates: First submitted 2023-01-22; First posted 2023-02-08 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Psychological Wellness; Resilience, Psychological; Personal and Professional Fulfilment; Wearable Devices; Multiomics
MeSH Terms: conditions — Psychological Well-Being | interventions — Chronology as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A subgroup of up to 300 participants will also undergo a microbiome sampling and will provide saliva and fasted blood samples at (see details below): (a) up to two weeks before DWD, as baseline; (b) at the end of the event. (c) one month after the event; (d) 3 months after the event; (e) 6 months after the event; (f) and one year after the event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DWD participants: Individuals that voluntarily chose to participate in DWD seminar.
  Interventions: Behavioral: Date With Destiny (DWD) Seminar
- Matched control group: Individuals that voluntarily chose to from the US population matched by gender, age, education, ethnicity and income

INTERVENTIONS:
Behavioral: Date With Destiny (DWD) Seminar — 6 days of immersive seminar
  Groups: DWD participants

SUMMARY:
The study approach is to leverage the most cutting-edge techniques of multi-omics biology, wearable physiology, and digital real-time psychology profiling and using machine learning models to understand the mechanisms underlying the strategies and techniques that enable participants the power to initiate and maintain sustainable behavior change.

Over the years, millions of people worldwide have attended immersive personal development seminars aiming to improve participants' health behaviors and wellness. Nevertheless, there's a scarcity of large-scale studies to assess their effects on behavior change and investigate their mechanism of action. A recent publication by the Science of Behavior Change Program (SOBC), launched by the National Institute of Health (NIH), recognized that: "science has not yet delivered a unified understanding of basic mechanisms of behavior change across a broad range of health-related behaviors, limiting progress in the development and translation of effective and efficacious behavioral intervention." As such, understanding the mechanisms underlying sustainable behavior change is key.

ELIGIBILITY:
Inclusion Criteria:

* 18-years-old and older
* English speaker
* Live in the US
* Participate in the DWD seminar (December 2-7, 2022)

Exclusion Criteria:

* Any physical or mental condition that limits the ability to participate in the study (e.g., answering e-questionnaires and wearing an electronic device)
* Serious active comorbidity or terminal illness
* Pregnancy
* Participation in any other clinical study focusing on psychological or behavioral intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals that voluntarily chose to participate in DWD seminar.
Sampling Method: Non-Probability Sample
Enrollment: 1445 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mental performance biomarker index. | one-year
  An algorithm will be used to create an index score using known biomarkers (psychosocial, physiological, and biological) related to participants' personalized mental performance. Higher index scores will indicate a better mental performance index. This outcome is assessed in the DWD group only.
Change from baseline in Oldenburg Burnout Inventory score (OLBI) | baseline through year one
  Participant self-report burnout assessed by OBLI survey, a 16-item questionarie assesing disengagement and exhaustion with a score range of 16-64, where higher scores indicate higher burnout; assessed in all participants.
Change from baseline in Percieved Stress Scale score (PSS-10) | baseline through year one
  Participant self-report perceived stress assessed by the Perceived Stress Scale (PSS-10), a 10-item questionnaire with a score range of 0-40, where higher scores indicate greater perceived stress; assessed in all participants.
Change from baseline in well-being score. | baseline through year one
  Participant self-report well-being assessed by the PERMA-H Profiler, a 23-item questionnaire measuring psychological well-being across five domains: positive and negative emotions, engagement, relationships, meaning, and accomplishment (range 0-10 per item, higher scores indicate greater well-being); assessed in all participants.
Change from baseline in subjective health score. | baseline through year one
  Participant self-report subjective health assessed by the health domain in the PERMA-H Profiler (range 0-10 per item, higher scores indicate higher subjective health); assessed in all participants.

SECONDARY OUTCOMES:
Change from baseline in Connor-Davidson Resilience Scale (CD-RISC-10) | baseline through year one
  Participant self-report resilience assessed by CD-RISC-10 survey, a 10-item questionarie assesing resilience with a score range of 0 - 40, where higher scores indicate greater resilience; assessed in all participants.
Change from baseline in General Self-Efficacy Scale (GSE-10) | baseline through year one
  Participant self-report self-efficacy assessed by GSE-10 survey, a 10-item questionarie assesing self-efficacy with a score range of 0 - 40, where higher scores indicate greater self-efficacy; assessed in all participants.
Change from baseline in Gratitude Questionnaire-Six Item Form (GQ-6) | baseline through year one
  Participant self-report gratitude assessed by the GQ-6 survey, a 6-item questionnaire measuring gratitude with a score range of 6-42, where higher scores indicate higher levels of gratitude; assessed in all participants.
Ecological Momentary Assessments (EMAs) score | baseline through year one
  EMAs scores rated by participants to assess momentary mood and cognitive states. This outcome is assessed in the DWD group only.
Professional Fulfillment Index (PFI) score | baseline through year one
  Participant self-report positive and negative facets of professional life assessed by PFI survey, a 16-item questionarie assesing fulfillment, work exhaustion, and interpersonal disengagement (range 0-4 per item). This outcome is assessed in the DWD group only.
WHO Quality of Life (WHO-QoL-BREF-26) score | baseline through year one
  Participant self-report quality of life assessed by the WHO-QoL-BREF-26 questionnaire, a 26-item questionnaire measuring physical health, psychological health, social relationships, and environmental health (each domain scored from 4 to 20, with higher scores indicating better quality of life). This outcome is assessed in the DWD arm only.
Growth-Fixed Mindset score | baseline through year one
  Participants self-report mindset assessed by the Growth and Fixed Mindset questionnaire, adapted to a 3-item questionnaire measuring growth/fixed mindset (higher scores indicating a stronger inclination toward a growth mindset). This outcome is assessed in DWD arm only.
Goals attainment score | baseline through year one
  Participant self-report goals attainment assessed by the goals achievement survey, a 14-item questionarie assessing participants' attainment of specific goals (range 0-10 per item). This outcome is assessed in the DWD group only.
Human Needs score | baseline through year one
  Participant self-report human needs assessed by the human needs survey, a 36-item questionnaire assessing participants' perceptions of their essential needs (range 0-10 per item). This outcome is assessed in the DWD group only.
Participants experiences and 0pinions | Up to 5 years after completion of the intervention
  Semi-structered Interviews with participants about their personal experiences and opinions after the workshop. This outcome will be assessed in DWD arm only.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Snyder, PhD, Principal Investigator — Stanford University; Shahar Lev-Ari, PhD, Principal Investigator — Stanford University & Tel-Aviv University
Locations (1):
- Stanford university, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding authors upon reasonable request. To protect participant privacy, individual-level data are not publicly available due to the sensitive nature of psychological and health-related information. Aggregated data and analysis scripts used to generate the main results and figures will be deposited in a public repository upon publication. Any additional data or materials required to replicate the reported findings that are not included in the public repository will be made available by the corresponding authors upon reasonable request, subject to institutional review board approval for sharing of de-identified data.